CLINICAL TRIAL: NCT02783053
Title: Metformin and Core Temperature in Obese and Lean Males
Acronym: McTOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: METC2015_117
Record Dates: First submitted 2015-10-19; First posted 2016-05-26 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin use (Other): The investigators compare the use of metformin vs no metformin
  Interventions: Drug: Metformin
- Lean or Obese (No Intervention): The investigators compare the effect of metformin on 18F-FDG uptake between lean and obese men.

INTERVENTIONS:
Drug: Metformin — Metformin vs no metformin
  Arms: Metformin use

SUMMARY:
Metformin is known to increase 18F-FDG uptake in subjects using metformin in retrospective trials.

In this study the researchers aim to investigate the influence of metformin (500 mg 1/day) on temperature in the colon, glucose uptake in the colon and energy expenditure in healthy lean (BMI < 24kg/m2) or obese subjects (BMI>28kg/m2). The investigators will measure 18F-FDG uptake in the colon, temperature in the colon, insulin sensitivity and energy expenditure before after using metformin.

DETAILED DESCRIPTION:
Obesity and diabetes mellitus type 2 (DM2) are health problems with a tremendous impact. Many attempts have been made to combat obesity and DM2, however, a breakthrough therapy is still lacking.

Obesity is the result of an imbalance between energy intake and energy expenditure. 18F-fluorodeoxy-d-glucose (18F-FDG) positron emission tomography computed tomography (PET-CT) pinpoint areas with high glucose turnover. Physiological 18F-FDG accumulation is frequently observed in the colon. Therefore, the colon might play an important role in increasing energy expenditure by consuming calories. However, the possibility of the colon as an energy dissipating tissue has not yet been explored. The colon could become an interesting new target of research to find a method to combat obesity.

Metformin is one of the few drugs in the treatment of DM2 that is associated with moderate weight loss. Interestingly, patients using metformin show an increased 18F-FDG-uptake in the colon. Whether this higher uptake of glucose also cause an increase in core temperature and/or an increase in energy expenditure is not known. The cause for this increase in glucose uptake in the colon by metformin use is unknown. Also, it is unknown whether this increase in glucose uptake results in an increased energy expenditure and/or an increase in core body temperature.

Objective: In this study the researchers aim to investigate the influence of metformin (500 mg 1/day) on temperature in the colon, glucose uptake in the colon and energy expenditure in healthy lean (BMI < 24kg/m2) or obese subjects (BMI>28kg/m2). The investigators will measure 18F-FDG uptake in the colon, temperature in the colon, insulin sensitivity and energy expenditure before after using metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian origin
* Subjects should be able and willing to give informed consent
* > 50 years old
* BMI< 24 kg/m2 or > 28 kg/m2

Exclusion Criteria:

* Renal failure (GFR< 60ml/min)
* Liver insufficiency (AST or alanine aminotransferase 3 times upper value)
* Chronic use of drugs or medication
* Diabetes mellitus
* Lactate acidosis or precoma diabeticum in medical history
* Acute or chronic diseases such as: dehydration, severe infection, shock, heartfailure, pulmonary insufficiency, recent heart attack
* Alcoholism

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
18F-FDG uptake | 1 week
  Difference in 18F-FDG uptake as registered by 18F-FDG PET-CT before and after 7 days of daily metformin use.

SECONDARY OUTCOMES:
Core temperature using a temperature pill | 48 hours
  - Difference in core body temperature before and after metformin
Correlation core temperature and 18F-FDG uptake | 1 week
  - Correlation between 18F-FDG uptake in the colon and core temperature
Energy expenditure (kcal/day) using ventilated hood | 30 minutes
  - Difference in energy expenditure before and after metformin use
Correlation between 18F-FDG uptake and energy expenditure | 1 week
  - Correlation between difference inenergy expenditure and 18F-FDG uptake in the colon

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands